CLINICAL TRIAL: NCT06966193
Title: Co-Producing LGBTQ-Affirmative Intervention Protocols for LGBTQ+ People at Risk of Self-Harm and Suicide: A Co-Production Study
Brief Title: Co-Producing LGBTQ-Affirmative DBT Protocols.
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Jake Camp, Adjunct Senior Lecturer, King's College London
Other Study IDs: 1072; NIHR304071 (Other Grant/Funding Number: National Institute of Health and Care Research)
Record Dates: First submitted 2025-04-24; First posted 2025-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Self-Harm; Suicidal; Emotional Dysregulation
Keywords: LGBTQ+; DBT; Self-Harm; Suicidal Behaviours; Emotion Dysregulation; Young People; Sexual Minorities; Gender Minorities; Co-Production; Adolescents; Therapists
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DBT Cohort Young Person Sample 1: Six to 12 young people who have completed at least four months of DBT, including those who did not complete the entire intended duration of the intervention or those still in the intervention, will be recruited via purposive sampling via the National & Specialist CAMHS DBT Service. If the investigators are unable to recruit sufficient numbers, they will seek to recruit from the adult DBT service within South London & Maudsley NHS Foundation Trust.
  Inclusion criteria will include that the young person:
  1. Is aged 13 to 21 years old;
  2. has completed at least four months of comprehensive DBT (i.e. inclusive of all four modes of intervention; Linehan, 1993; Miller et al., 2006; Rathus & Miller, 2015) in the past 24 months or have completed at least four months of DBT and are still in a comprehensive DBT programme;
  3. identifies as LGBTQ+ (including those questioning or unsure about their orientation/identity);
  4. is willing and able to participate in the study.
- Non-DBT Cohort Young Person Sample 2: Six to 12 young people who have experienced difficulties with at least one of the identified intervention targets (identity confusion, managing stigma experiences, and connecting with similar others) will be recruited from CAMHS and from community organisations (e.g. LGBTQ+ charities).
  Inclusion criteria will follow similar to sample 1. The young person:
  1. Is aged 13 to 21 years old;
  2. has not accessed and is not currently enrolled in a comprehensive DBT programme;
  3. has experienced difficulties with LGBTQ-related identity confusion, managing stigma experiences, and connecting with similar others;
  4. identifies as LGBTQ+ (including those questioning or unsure about their orientation/identity);
  5. is willing and able to participate in the study (i.e. are based in the UK and can attend the in-person and online groups).
- DBT Therapist Sample: Four to eight DBT therapists will be recruited via purposive sampling via the National & Specialist CAMHS DBT Service and Adult DBT Services in South London & Maudsley NHS Foundation Trust. Inclusion criteria will include:
  1. Currently practicing or having completed (or recently finished, within the past 12 months) a comprehensive DBT programme as a DBT therapist. In order to practice as a DBT therapist, they must hold a professional qualification recognised by appropriate healthcare regulators.
  2. Having experience working with at least one LGBTQ+ client in DBT, who was aged between 13 and 21 years at the time.
  3. Being willing and able to participate in the study.

SUMMARY:
Aims:

1. To co-produce new intervention parts that meet the needs of LGBTQ+ people at risk of self-harm or suicidal thoughts, with LGBTQ+ people and DBT therapists. These intervention parts will be integrated into a Dialectical Behaviour Therapy (DBT) intervention, that is provided earlier in a persons mental health care journey, than DBT is usually targeted at.
2. To assess how acceptable and feasible the co-production process was for participants, and how well it achieved co-production principles (e.g. participants feel supported, that the aims were transparent, etc).

Why is This Important? Young people who identify as lesbian, gay, bisexual, transgender, queer, and with other minoritised gender and sexual identities (LGBTQ+) are much more likely to self-harm and experience suicidal thoughts than cisgender-heterosexual (non-LGBTQ+) people. They also experience barriers when accessing mental health support. Some of these barriers come from a lack of support tailored towards their needs as an LGBTQ+ person. This often means that things get worse before they access the right support, and so are often seen in higher-intensity interventions (tier 4 or tertiary care), like DBT.

What The Investigators Plan to Do:

The investigators plan to hold some focus groups with three different groups of people to co-produce the new intervention parts. The three groups include:

1. A group of LGBTQ+ young people (13-21 years old) who have completed a at full DBT programme recently.
2. A group of LGBTQ+ young people (13-21 years old) who have never been in a full DBT programme but experienced similar difficulties.
3. A group of DBT therapists who have supported LGBTQ+ young people before.

The investigators will seek feedback from participants about how acceptable they found the study (e.g. how satisfied they were with the process), how feasible it was (e.g. were they able to attend and was it practice?), and how well they stuck to the coproduction principles (e.g. how supported they felt).

ELIGIBILITY:
DBT Cohort Young Person Sample 1

Inclusion criteria will include that the young person:

1. Is aged 13 to 21 years old;
2. has completed at least four months of comprehensive DBT (i.e. inclusive of all four modes of intervention; Linehan, 1993; Miller et al., 2006; Rathus & Miller, 2015) in the past 24 months or have completed at least four months of DBT and are still in a comprehensive DBT programme;
3. identifies as LGBTQ+ (including those questioning or unsure about their orientation/identity);
4. is willing and able to participate in the study. While no specific inclusion or exclusion criteria will be placed on other variables, typically to be eligible for a DBT programme, young people would need to have a history of self-harm and/or suicidal behaviours, difficulties with emotion regulation, and potentially difficulties with the remaining symptom list within borderline/emotionally unstable personality disorder. Recruitment size is based on PPI recommendations regarding effective group sizes, with allowances for sample attrition.

Non-DBT Cohort Young Person Sample 2

Inclusion criteria will follow similar to sample 1. The young person:

1. Is aged 13 to 21 years old;
2. has not accessed and is not currently enrolled in a comprehensive DBT programme;
3. has experienced difficulties with LGBTQ-related identity confusion, managing stigma experiences, and connecting with similar others;
4. identifies as LGBTQ+ (including those questioning or unsure about their orientation/identity);
5. is willing and able to participate in the study (i.e. are based in the UK and can attend the in-person and online groups).

No other inclusion or exclusion criteria will be systematically implemented for this group.

DBT Therapist Sample

Inclusion criteria:

1. Currently practicing or having completed (or recently finished, within the past 12 months) a comprehensive DBT programme as a DBT therapist. In order to practice as a DBT therapist, they must hold a professional qualification recognised by appropriate healthcare regulators.
2. Having experience working with at least one LGBTQ+ client in DBT, who was aged between 13 and 21 years at the time.
3. Being willing and able to participate in the study.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: DBT Cohort Young Person Sample 1 Young people will be recruited via purposive sampling via the National & Specialist CAMHS DBT Service and the adult DBT service within South London & Maudsley NHS Foundation Trust.
  Non-DBT Cohort Young Person Sample 2 Young people will be recruited from CAMHS within South London & Maudsley NHS Foundation Trust and from community organisations (e.g. LGBTQ+ charities) and general advertising on social media and similar.
  DBT Therapists DBT therapists will be recruited via purposive sampling via the National & Specialist CAMHS DBT Service and Adult DBT Services in South London & Maudsley NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility/Recruitment | Baseline
  Whether the investigators are able to recruit the intended numbers of participants to each group by the start of the focus groups (baseline).
Feasibility/Attrition | Baseline, during the focus groups (12 weeks in duration), and at outcome measure completion (12 weeks from baseline)
  Participant attrition rates at baseline, during the study, and at outcome measure completion (12 weeks from baseline).
Feasibility/Focus Group Content and Delivery | For the duration of the focus groups (12 weeks)
  The count frequency of focus groups, individual sessions, and duration of each taken will be recorded. The content of the focus groups will be documented. The number of facilitators of each type will also be documented.
Acceptability/Session Satisfaction | At the end of each focus group (6 focus groups over 12 weeks)
  Self-report question at the end of each focus group/individual session: How satisfied were you with the focus group/individual session? [Response Options: Very Satisfied, Satisfied, Neutral, Unsatisfied, Very Unsatisfied].
  [Prompt] Can you tell us why you gave that rating? [Prompt] what would have improved your satisfaction?
Acceptability/Satisfaction with the Study | End of Study (12 weeks post baseline)
  End of study feedback:
  How satisfied were you with the focus group/individual sessions overall? Response Options: Very Satisfied, Satisfied, Neutral, Unsatisfied, Very Unsatisfied. Prompts to elicit qualitative feedback.
  How satisfied were you with the final version of the intervention protocols that we all produced together? Response Options: Very Satisfied, Satisfied, Neutral, Unsatisfied, Very Unsatisfied. Prompts to elicit qualitative feedback.
Acceptability/Recommend to Others | End of study (12 weeks post baseline)
  End of study feedback:
  Would you recommend this study to other potential LGBTQ+ people if we were to run the study again? [Response Options] Yes, No, Maybe [Prompt] Can you tell us why you gave that rating?
Acceptability/Helpfulness | End of study (12 weeks post baseline)
  End of study feedback:
  Did you find participating in this study helpful to you? [Response Options] Yes, No, Maybe [Prompt] Can you tell us why you have that rating? [Prompt] What would have made it more useful?
Acceptability/Engagement | End of study (12 weeks post baseline)
  End of study feedback:
  [Acceptability/Engagement.] What helped you to engage in the focus groups?[Acceptability/Engagement.] What got in the way of engaging in the focus groups?
Acceptability/Cultural Sensitivity | End of study (12 weeks post baseline)
  End of study Feedback:
  [Acceptability/Cultural Sensitivity.] Did the content of the focus groups feel respectful and relevant for LGBTQ+ culture and potential intersecting cultures within the community? [Response Options] Yes, No, Maybe [Prompt] Can you tell us why you gave that rating? [Prompt] Were there any blind spots in this regard? [Prompt] What could we have done differently to improve respect and relevance? [Prompt] What worked well in this regard?
Feasibility/General | End of study (12 weeks post baseline)
  End of study feedback:
  How feasible was it for you to take part in this project? [Prompt] Feasible means how possible it was to do this easily or conveniently. [Response Options] Very Feasible, Feasible, Neither Feasible or Unfeasible, Unfeasible, Very Unfeasible [Prompt] Can you tell us why you gave that rating? [Prompt] What made it more feasible? [Prompt] What were the barriers to it being feasible?
Feasibility/Practicalities | End of study (12 weeks post baseline)
  End of study feedback:
  [Feasibility/Practicality.] Can you tell us how you found the practicalities of the workshop, including but not limited to the timings, the environment they were conducted in (online vs in-person), the types of activities used, and so forth? [Prompt] cover any in the list which the participant did not speak to [Prompt] How did this impact the feasibility of taking part, if at all? [Prompt] What would you recommend to improve any future similar studies in regards to practicalities?

SECONDARY OUTCOMES:
Wellbeing | End of study (12 weeks post baseline)
  End of study feedback:
  [Wellbeing.] Did taking part in this project have any impact on your wellbeing? This can be positive, negative, or neutral?
Co-Production Process/Respect | End of study (12 weeks post baseline)
  My contributions within the whole study felt respected and acknowledged. [Response Options: Very True, True, Neutral, Untrue, Very Untrue]. [Prompt] Can you tell us why? [Prompt] What worked well? [Prompt] What worked less well? [Prompt] Recommendations for improving this?
Co-Production Process/Support | End of study (12 weeks post baseline)
  I felt adequately supported within the whole study (e.g. my expenses were covered, I was offered support if needed, my questions were answered, etc).
  [Response Options: Very True, True, Neutral, Untrue, Very Untrue]. [Prompt] Can you tell us why? [Prompt] What made you feel supported? [Prompt] What didn't make you feel supported? [Prompt] Recommendations for improving this?
Co-production Process/Transparency | End of study (12 weeks post baseline)
  The aims of the study and of my involvement were clear to me. [Response Options: Very True, True, Neutral, Untrue, Very Untrue] [Prompt] Can you tell us why? [Prompt] What worked well? [Prompt] What worked less well? [Prompt] Recommendations for improving this?
Co-Production Process/Responsiveness | End of study (12 weeks post baseline)
  I felt listened to and like my contributions were responded to in the study. [Response Options: Very True, True, Neutral, Untrue, Very Untrue]. [Prompt] Can you tell us why? [Prompt] What worked well? [Prompt] What worked less well? [Prompt] Recommendations for improving this?
Co-Production Process/Fairness of Opportunities | End of study (12 weeks post baseline)
  I felt like everyone was given fair opportunities, especially in the context of diversity within the group? [Response Options: Very True, True, Neutral, Untrue, Very Untrue]. [Prompt] Can you tell us why? [Prompt] What worked well? [Prompt] What worked less well? [Prompt] Recommendations for improving this?
Co-production Process/Accountability | End of study (12 weeks post baseline)
  I felt accountable for my involvement in the study and was able to provide feedback.
  [Response Options: Very True, True, Neutral, Untrue, Very Untrue]. [Prompt] Can you tell us why? [Prompt] What worked well? [Prompt] What worked less well? [Prompt] Recommendations for improving this?
Co-Production/Empowerment | End of study (12 weeks post baseline)
  Did you feel empowered to take part in the study? [Response Options: Very True, True, Neutral, Untrue, Very Untrue]. [Prompt] Can you tell us why? [Prompt] What worked well? [Prompt] What worked less well? [Prompt] Recommendations for improving this?

IPD SHARING:
Plan to Share IPD: No
The majority of the data is qualitative and thus would have cause problems with anonymity if IPD was made available.